CLINICAL TRIAL: NCT01839526
Title: A Cross-sectional Study of Renal Function in Treatment-naïve, Young Male Patients With Fabry Disease
Brief Title: A Study of Renal Function in Treatment-naïve, Young Male Patients With Fabry Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment period not extended and screening stopped for slow recruitment and in accordance with provisions of the protocol. Not linked to any safety concern
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGAL19110; 2012-001966-14 (EudraCT Number); MSC 12711 (Other: Sanofi)
Record Dates: First submitted 2013-04-11; First posted 2013-04-25 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2016-10

CONDITIONS: Fabry Disease
Keywords: Fabry disease
MeSH Terms: conditions — Fabry Disease | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glomerular Filtration Rate by Plasma Iohexol Clearance (iGFR) (Other): Evaluations of renal and cardiac function
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Evaluations of renal and cardiac function are standard-of-care in young patients with Fabry disease. This study uses the more precise iGFR measurement of renal function. No investigational drug will be administered in this study for the treatment of Fabry disease.

SUMMARY:
No investigational drug will be administered in this study for the treatment of Fabry disease.

This will be a multicenter, multinational, non-treatment, cross-sectional study of young male patients with Fabry disease who have not yet initiated interventional treatment for this disease. The study will consist of a screening visit(s), a clinical investigation visit(s), and a follow-up phone contact.

The objectives of the study are:

* To document renal function and other Fabry disease manifestations across age in treatment-naïve, young male patients with Fabry disease.
* To provide a reference group for comparison with interventional clinical trials of Fabry disease.

The duration of each patient's participation in the study, inclusive of the screening visit and follow-up phone contact, will be approximately 12 weeks.

DETAILED DESCRIPTION:
Patients who meet all eligibility criteria based on screening assessments will be scheduled to return to the clinic for assessments of renal function and other disease-related parameters, which may be scheduled over one or more clinical investigation visits. The clinical investigation visit(s) will be scheduled such that renal and cardiac assessments occur after the required medication washout (see exclusion criterion); other procedures may be performed either before or after the medication washout, at the discretion of the investigator.

Up to 100 patients will be enrolled in the study, including a minimum of 15 patients in each of the following age groups (based on age at screening): 5 to 11 years, 12 to 17 years, and 18 to 25 years.

All patients will be encouraged to enroll in the Fabry Registry (NCT00196742) for continued follow-up after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient and/or their parent/legal guardian is willing and able to provide signed informed consent. If the patient is below the age of consent per local guidelines, he is willing to provide assent, if deemed able to do so.
* The patient must have a confirmed diagnosis of Fabry disease as documented by leukocyte α-galactosidase A (αGAL) of <4 nmol/hr/mg leukocyte (preferred assay; results from a central laboratory). If the leukocyte αGAL activity assay is difficult to obtain, the patient may be enrolled based on documented plasma αGAL <1.5 nmol/hr/mL (results from a central laboratory), with the agreement of the Genzyme Medical Monitor.

Exclusion Criteria:

* Patient has received prior treatment with enzyme replacement therapy (ERT) or oral pharmacological chaperone therapy for Fabry disease.
* Patient has received an investigational drug within 30 days of the screening visit.
* Patient is receiving any of the following medications and is clinically unable or unwilling to temporarily discontinue treatment with these medications for the indicated washout period prior to the renal function assessments until completion of these assessments:

  * Angiotensin converting enzyme inhibitors or angiotensin receptor blockers (6 week washout);
  * Non-steroidal anti-inflammatory drugs (3 day washout).
  * NOTE: Patients who are on chronic dialysis or have had a kidney transplant will not be required to discontinue the above medications because renal function assessments will not be performed in these patients.
* Patient has any contraindication mentioned in the labeling of iohexol. NOTE: patients with an eGFR <30 mL/min/1.73m^2 and patients who are on chronic dialysis or have had a kidney transplant may be enrolled irrespective of any contraindication to iohexol because iGFR will not be measured in these patients.
* Patient has any medical condition or extenuating circumstance which, in the opinion of the Investigator, could interfere with the patient's ability to complete all study procedures, or with the interpretation of study results (e.g., diabetes mellitus).
* The patient and/or their parent or legal guardian, in the opinion of the Investigator, is unable to adhere to the requirements of the study.

Ages: 5 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate Estimated from Serum Creatinine (eGFR) | Day 1 to Week 8
  Tests are performed only for patients who are not on chronic dialysis and/or have not received a kidney transplant.
Glomerular Filtration Rate by Plasma Iohexol Clearance (iGFR) | Day 1 to Week 8
  Assessment of iGFR will NOT be performed if a patient is on chronic dialysis, has had a kidney transplant, or has a screening eGFR <30 mL/min/1.73 m^2 or presents any contraindication mentioned in the labeling of iohexol (Omnipaque™ 300).
Protein Excretion Assessed from Three First-Morning Urine Voids | Day 1 to Week 12

SECONDARY OUTCOMES:
Cardiovascular Function | Day 1 to Week 8
  Assessed by electrocardiogram (ECG) and echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (22):
- United States (5):
  - Investigational Site Number 840010, La Jolla, California
  - Investigational Site Number 840006, Decatur, Georgia
  - Investigational Site Number 840003, Cincinnati, Ohio
  - Investigational Site Number 840009, Salt Lake City, Utah
  - Investigational Site Number 840002, Fairfax, Virginia
- Investigational Site Number 032001, Capital Federal, Argentina
- Investigational Site Number 040001, Vienna, Austria
- Investigational Site Number 056001, Liège, Belgium
- Investigational Site Number 076001, Porto Alegre, Brazil
- Canada (2):
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124004, Toronto
- Investigational Site Number 246002, Vaasa, Finland
- France (2):
  - Investigational Site Number 250002, Bron
  - Investigational Site Number 250001, Garches
- Investigational Site Number 348001, Pécs, Hungary
- Investigational Site Number 578001, Bergen, Norway
- Investigational Site Number 616001, Warsaw, Poland
- Spain (2):
  - Investigational Site Number 724001, Badalona
  - Investigational Site Number 724002, Girona
- Investigational Site Number 158001, Taipai, Taiwan
- United Kingdom (2):
  - Investigational Site Number 826004, London
  - Investigational Site Number 826002, London